CLINICAL TRIAL: NCT05882903
Title: The Effect of Intra-sinus Application of Betamethasone Dipropionate Nasal Cream on Patients with Chronic Rhinosinusitis Post Functional Endoscopic Sinus Surgery (FESS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oticara Australia PTY LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OT-007B
Record Dates: First submitted 2023-05-12; First posted 2023-05-31 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Betamethasone Dipropionate Nasal Cream 0.0644% Treatment (Experimental): Betamethasone Dipropionate Nasal Cream 0.0644% is applied topically to the inflamed tissue of the sinus using a pre-filled syringe and applicator under the guidance of an endoscope. Up to 5g on each side of the sinus (10g in total).
  Interventions: Drug: Betamethasone Dipropionate Nasal Cream 0.0644%; Device: Pre-filled syringe and applicator device

INTERVENTIONS:
Drug: Betamethasone Dipropionate Nasal Cream 0.0644% — Betamethasone Dipropionate Nasal Cream 0.0644% is applied topically to the inflamed tissue of the sinus using a pre-filled syringe and applicator under the guidance of an endoscope. Up to 5g on each side of the sinus (10g in total).
Device: Pre-filled syringe and applicator device — Cream is pre-filled to a syringe and applicator device to facilitate the topical application direct to the sinus under endoscopic guidance.

SUMMARY:
To assess the safety and efficacy of one (single) application of Betamethasone Dipropionate Nasal Cream (BMDP CREAM) onto the sinus mucosa.

DETAILED DESCRIPTION:
In this open-label study, a single dose of the corticosteroid Betamethasone Dipropionate Nasal Cream 0.0644% (equivalent to 0.05% Betamethasone) will be administered under endoscopic guidance to the sinus mucosa of post-FESS patients whose chronic rhinosinusitis (CRS) condition is suboptimal under the current standard of care. The safety and benefits of this treatment will be monitored by patient-reported symptoms and endoscopic assessment of the sinus mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a clinically confirmed diagnosis of CRS by an otolaryngologist (ENT) undergoing maximal medical therapy as part of their standard of care.
* Having undergone functional endoscopic sinus surgery (FESS) at least 6 months prior to enrolment.
* For each nostril, an endoscopic nasal polyp score of 0, 1, or 2 out of a maximum score of - (where 0= No polyps, 1= small polyps in the middle meatus not reaching below the inferior border of the middle turbinate , 2= nasal polyps reaching below the border of the middle turbinate, 3= large nasal polyps reaching the lower border of the inferior turbinate or nasal polyps medial to the middle turbinate, 4= large nasal polyps causing almost complete obstruction of the inferior nasal cavity) (Gevaert et al, 2023).
* Visible middle turbinates and access to the ethmoid sinuses for dosing as established via endoscopic examination.
* Participants must have a > 2 on the disease severity visual analogue scale (VAS) at screening and pre-treatment.
* Body weight: A minimum body weight >=40 kilograms (kg) and a BMI of ≤ 39 at the screening visit.
* Individuals of childbearing potential must use adequate birth control methods and not plan to get pregnant during the study.
* Informed consent: Willingness to give written informed consent and willingness to participate in and comply with the study.
* Age ≥18 but <80 years.

Exclusion Criteria:

* Subjects with known hypersensitivity or contraindications to betamethasone dipropionate, mometasone, or topical anaesthesia.
* Subjects with sino-nasal abnormalities, disease, or implanted devices that prevents the application of the therapy.
* Previous enrolment in this study.
* Subjects currently receiving systemic corticosteroid or have received systemic corticosteroid in the prior 4 weeks or receiving biologic therapy.
* Subjects with a history of glaucoma or cataracts or have an abnormal intraocular pressure (IOP) at screening or pre-treatment (abnormal IOP is defined as greater than 21 mm Hg).
* Subjects with acute sinusitis.
* Subjects with known immunodeficiency.
* Subjects with diabetes (Type 1).
* Subjects with cystic fibrosis.
* Pregnant subjects or subjects trying to get pregnant or currently lactating as the effect on human pregnancy is unknown.
* Subjects who are unable to give an informed consent because of mental illness, dementia or communication difficulties.
* Subjects with a Cushing's disease diagnosis within the previous 12 months.
* Severe septal deviation and or previous total resection of the middle turbinate.
* Any lab abnormality or underlying medical condition which, in the Investigator's opinion, should exclude the participant.
* Subjects who are unlikely to comply with study procedures, restrictions and requirements as determined by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in 4-Cardinal Symptom score (4CSS) Baseline to Week 3. | Baseline through study completion, an average of 4 weeks
  Change in average daily score prior to dosing (an average of 7 days) and the average daily score of the 7 days prior to exit (between week 2 and 3 weeks after dosing).Participants score their 4-Cardinal Symptom score (4CSS) daily on a Likert scale of 0-5; where 0= no problem - 5= problem as bad as can be, higher scores indicate higher severity of symptoms.
Change in SNOT-22 Baseline to Week 3. | Baseline through study completion, an average of 4 weeks
  Participants complete the Sino-nasal Outcome Test (SNOT-22) questionnaire at Baseline and Week 3, analysis will focus on the nasal symptom subdomain. The SNOT-22 measures 22 symptoms on a Likert scale of 0-5; where 0= no problem - 5= problem as bad as can be, higher scores indicate higher severity of symptoms. A higher total score indicates greater symptom severity.

SECONDARY OUTCOMES:
Safety of one application of BMDP Cream onto the sinus mucosa. | Informed consent through study completion, an average of 3 weeks
  Monitoring of morning serum cortisol levels, glucose levels, treatment emergent changes in other chemistry or haematology results deemed clinically significant by the Investigator, intraocular pressure, and BMDP Cream application related adverse events.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Oticara Investigational Site, Sydney, New South Wales
  - Oticara Investigational Site, Brisbane, Queensland
  - Oticara Investigational Site, Adelaide, South Australia
  - Oticara Investigational Site, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No